CLINICAL TRIAL: NCT00004096
Title: A Phase I/II Study of Carboplatin and Navelbine for Advanced Non-Small Cell Lung Cancer
Brief Title: Carboplatin Plus Vinorelbine in Treating Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 99L2; NU-99L2; NCI-G99-1589
Record Dates: First submitted 1999-12-10; First posted 2004-08-05 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: carboplatin
Drug: vinorelbine ditartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining carboplatin and vinorelbine in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility of chemotherapy with carboplatin and vinorelbine in patients with stage IIIB or IV non-small cell lung cancer. II. Determine the maximum tolerated dose and dose limiting toxicities of this regimen in these patients. III. Determine the response rate and survival of these patients after this treatment.

OUTLINE: This is a dose escalation study of vinorelbine. Patients receive carboplatin IV over 30 minutes followed by vinorelbine IV over 6-10 minutes on days 1 and 8. Treatment repeats every 21 days in the absence of unacceptable toxicity or disease progression. Cohorts of 3-6 patients receive escalating doses of vinorelbine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 2 of 6 patients experience dose limiting toxicity. Patients are followed at 1 month.

PROJECTED ACCRUAL: A total of 12-36 patients will be accrued for this study over 6-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven stage IIIB or IV non-small cell lung cancer

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 8 weeks Hematopoietic: WBC at least 3000/mm3 Absolute neutrophil count at least 1500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal SGOT no greater than 3 times normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 50 mL/min Other: No significant active infection No other severe medical illness No prior significant symptomatic peripheral neuropathy (grade 2 or worse) No concurrent neuropathy Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 3 weeks since prior chemotherapy and recovered No more than 1 prior chemotherapy regimen No prior vinorelbine Endocrine therapy: Not specified Radiotherapy: Recovered from any prior radiotherapy No prior radiotherapy to more than 10% of bone marrow Surgery: At least 2 weeks since prior major surgery and recovered Other: At least 30 days since prior experimental therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A. Masters, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States